CLINICAL TRIAL: NCT00281931
Title: Phase II Trial of Combined Immunochemotherapy With Fludarabine, Cyclophosphamide and Rituximab in Patients With B-PLL
Brief Title: Fludarabine, Cyclophosphamide, and Rituximab in Treating Patients With Prolymphocytic Leukemia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: German CLL Study Group (Other)
Allocation: Non-Randomized | Masking: None | Purpose: Treatment
Other Study IDs: PLL1; EU-20563
Record Dates: First submitted 2006-01-24; First posted 2006-01-25 (Estimated); Last update posted 2016-09-26 (Estimated); Status verified 2016-09

CONDITIONS: Prolymphocytic Leukemia
Keywords: prolymphocytic leukemia
MeSH Terms: conditions — Leukemia, Prolymphocytic | interventions — Rituximab; Cyclophosphamide; fludarabine phosphate

INTERVENTIONS:
Biological: rituximab
Drug: cyclophosphamide
Drug: fludarabine phosphate

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as fludarabine and cyclophosphamide, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as rituximab, can block cancer growth in different ways. Some find cancer cells and kill them or carry cancer-killing substances to them. Others interfere with the ability of cancer cells to grow and spread. Giving fludarabine and cyclophosphamide together with rituximab may kill more cancer cells.

PURPOSE: This phase II trial is studying how well giving fludarabine and cyclophosphamide together with rituximab works in treating patients with B-cell prolymphocytic leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the overall and progression-free survival of patients with B-cell prolymphocytic leukemia treated with immunochemotherapy comprising fludarabine, cyclophosphamide, and rituximab.
* Determine the toxic effects of this regimen in these patients.

OUTLINE: This is a non-randomized, open-label, multicenter study.

Patients receive fludarabine IV and cyclophosphamide IV on days 1-3. Patients also receive rituximab IV on day 0 in course 1 and on day 1 in courses 2-6. Treatment repeats every 28 days for up to 6 courses.

PROJECTED ACCRUAL: A total of 21 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of B-cell prolymphocytic leukemia

  * Previously treated disease
* All Binet stages allowed

PATIENT CHARACTERISTICS:

* Life expectancy > 3 months
* ECOG/WHO performance status 0-3

PRIOR CONCURRENT THERAPY:

* No more than 3 prior treatment regimens

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 1999-09; Primary Completion 2006-04 (Actual); Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Overall survival
Progression-free survival
Toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Michael Herold, MD, PhD, Study Chair — HELIOS Hospital, Erfurt, Germany
Locations (1):
- Helios Klinikum Erfurt, Erfurt, Germany

IPD SHARING:
Plan to Share IPD: No